CLINICAL TRIAL: NCT02687191
Title: A PHASE 1B MULTICENTER, OPEN-LABEL STUDY TO EVALUATE THE SAFETY AND TOLERABILITY AND DETERMINE THE MAXIMUM TOLERATED DOSE OF PF-05230907 IN SUBJECTS WITH INTRACEREBRAL HEMORRHAGE (ICH)
Brief Title: Safety and Tolerability of PF-05230907 in Intracerebral Hemorrhage
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: B2341002 was terminated on 26-OCT-2017 for strategic reasons. The decision to terminate the trial was not based on any safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2341002; 2015-005703-83 (EudraCT Number)
Record Dates: First submitted 2016-02-16; First posted 2016-02-22 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Intracerebral Hemorrhage
Keywords: safety, maximum tolerated dose, modified continual reassessment method, intracerebral, hemorrhage, hematoma
MeSH Terms: conditions — Cerebral Hemorrhage; Hemorrhage; Hematoma | interventions — PF-05230907

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- PF-05230907 (Cohort 1) (Experimental): PF-05230907 IV bolus injection
  Interventions: Biological: PF-05230907
- PF-05230907 (Cohort 2) (Experimental): PF-05230907 IV bolus injection
  Interventions: Biological: PF-05230907
- PF-05230907 (Cohort 3) (Experimental): PF-05230907 IV bolus injection
  Interventions: Biological: PF-05230907
- PF-05230907 (Cohort 4) (Experimental): PF-05230907 IV bolus injection
  Interventions: Biological: PF-05230907
- PF-05230907 (Cohort 5) (Experimental): PF-05230907 IV bolus injection
  Interventions: Biological: PF-05230907
- PF-05230907 (Cohort 6) (Experimental): PF-05230907 IV bolus injection
  Interventions: Biological: PF-05230907
- PF-05230907 (Cohort 7) (Experimental): PF-05230907 IV bolus injection
  Interventions: Biological: PF-05230907
- PF-05230907 (Cohort 8) (Experimental): PF-05230907 IV bolus injection
  Interventions: Biological: PF-05230907
- PF-05230907 (Cohort 9) (Experimental): PF-05230907 IV bolus injection
  Interventions: Biological: PF-05230907
- PF-05230907 (Cohort 10) (Experimental): PF-05230907 IV bolus injection
  Interventions: Biological: PF-05230907
- PF-05230907 (Cohort 11) (Experimental): PF-05230907 IV bolus injection
  Interventions: Biological: PF-05230907
- PF-05230907 (Cohort 12) (Experimental): PF-05230907 IV bolus injection
  Interventions: Biological: PF-05230907
- PF-05230907 (Cohort 13) (Experimental): PF-05230907 IV bolus injection
  Interventions: Biological: PF-05230907
- PF-05230907 (Cohort 14) (Experimental): PF-05230907 IV bolus injection
  Interventions: Biological: PF-05230907
- PF-05230907 (Cohort 15) (Experimental): PF-05230907 IV bolus injection
  Interventions: Biological: PF-05230907

INTERVENTIONS:
Biological: PF-05230907 — PF-05230907 IV bolus injection

SUMMARY:
This study employs a modified continual reassessment method (mCRM) design to estimate the maximum tolerated dose (MTD) of PF-05230907, defined as a target toxicity rate of 15% based on treatment emergent thromboembolic and/or ischemic events (TIEs). The mCRM design utilizes Bayesian methodology to continuously learn the dose-toxicity relationship, which is characterized by a parametric model.

Subjects with a diagnosis of ICH (determined by computed tomography) will be enrolled in cohorts of 3. The total length of time planned for study participation is approximately 3 months; 6.0 hours for screening, a single dose administration with a 4-day minimum hospital confinement period and follow-up visits through Day 91.

Severity of adverse events (AEs) and serious adverse events (SAEs) will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. All subjects who receive PF-05230907 are evaluable for TIEs. The determination of MTD using mCRM modeling will be based on TIEs which occur through 7 days post-dose (Day 8).

ELIGIBILITY:
Inclusion Criteria:

* ICH as documented by CT scan within 6.0 hours of symptom onset
* Baseline ICH volume > 5mL and < 60 mL

Exclusion Criteria:

* Deep coma (Glasgow Coma Scale < 6)
* Modified Rankin Score > 3 prior to ICH onset
* Known history of schemic, vaso-occlusive or thrombotic events within 6 months prior to screening
* Known prothrombotic disorders
* Known secondary ICH related to aneurysm, arteriovenous malformation, subarachnoid hemorrhage, trauma, or other causes. CT angiography, MR, or other diagnostic studies obtained as part of the standard of care may be used to assess eligibility.
* Known use of oral anticoagulant(s)
* Known use of low-molecular weight heparin or heparin

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- United States (5):
  - Barnes Jewish Hospital, St Louis, Missouri
  - Washington University,, St Louis, Missouri
  - James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Martha Morehouse Medical Plaza, Columbus, Ohio
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- Spain (5):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clínico Universitario de Santiago de Compostela, Area Neurovascular-Neurologia, Santiago de Compostela, LA Coruna
  - Hospital Vall d'Hebron, Unidad de Ictus, Barcelona
  - Hospital Universitari Dr. Josep Trueta IDIBGI, Department Neurology, Girona
  - Hospital Universitario Ramon y Cajal, Madrid
- University College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Silva Blas Y, Diringer MN, Lo B, Masjuan J, Perez de la Ossa N, Cardinal M, Yong F, Zhu T, Li G, Arkin S. Phase 1b Study to Evaluate Safety, Tolerability, and Maximum Tolerated Dose of PF-05230907 for Intracerebral Hemorrhage. Stroke. 2021 Jan;52(1):294-298. doi: 10.1161/STROKEAHA.120.029789. Epub 2020 Dec 4. PMID 33272131
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2341002&StudyName=A%20Phase%201b%20Multicenter%2C%20Open-label%20Study%20To%20Evaluate%20The%20Safety%20And%20Tolerability%20To%20Determine%20The%20Maximum%20Tolerated%20Dose%20Of%20Pf-05230907%20In%20Intracerebral%20Hemorrhage%20%28ich%29%20Subjects
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2341002&StudyName=A+Phase+1b+Multicenter%2C+Open-label+Study+To+Evaluate+The+Safety+And+Tolerability+And+Determine+The+Maximum+Tolerated+Dose+Of+Pf-05230907+In+Subjects+With+Intracerebral+Hemorrhage+%28ich%29

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Not all the 15 pre-specified dose groups (possible doses based on Bayesian modified continual reassessment method [mCRM]) were expected to be studied. The actual doses were determined by mCRM and safety review. Study results were reported for the 6 actual dose groups allocated with participants.
Groups:
- PF-05230907 5 Microgram Per Kilogram (mcg/kg): PF-05230907 5 mcg/kg was administered as a single intravenous (IV) bolus on Day 1.
- PF-05230907 8 mcg/kg: PF-05230907 8 mcg/kg was administered as a single IV bolus on Day 1.
- PF-05230907 12 mcg/kg: PF-05230907 12 mcg/kg was administered as a single IV bolus on Day 1.
- PF-05230907 19 mcg/kg: PF-05230907 19 mcg/kg was administered as a single IV bolus on Day 1.
- PF-05230907 24 mcg/kg: PF-05230907 24 mcg/kg was administered as a single IV bolus on Day 1.
- PF-05230907 30 mcg/kg: PF-05230907 30 mcg/kg was administered as a single IV bolus on Day 1.
Period: Overall Study
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Started | 3 | 3 | 3 | 6 | 3 | 3
Completed | 3 | 2 | 2 | 5 | 2 | 2
Not Completed | 0 | 1 | 1 | 1 | 1 | 1
Not completed — Death | 0 | 1 | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received the treatment of PF-05230907.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (5.5) | 65.7 (5.5) | 62.3 (11.9) | 62.2 (8.1) | 66.7 (3.8) | 67.7 (9.6) | 62.3 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2 | 1 | 0 | 2 | 7
  Male | 1 | 3 | 1 | 5 | 3 | 1 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 3 | 3 | 4 | 3 | 3 | 18
  Black | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Thromboembolic and/or Ischemic Events (TIEs)
Description: Thromboembolic and/or ischemic events (TIEs) were defined as any of the following events: disseminated intravascular coagulation (Grade [Gr]>=3); acute coronary syndrome (Gr >=3); cardiac arrest (Gr >=4); myocardial infarction (Gr >=3); Cardiac troponin I increased (Gr 3); ischemia cerebrovascular (Gr >=1 and associated with lesion[s]); portal vein thrombosis (Gr >=2); ischemic stroke (Gr >=1 and associated with lesion[s]); transient ischemic attacks (Gr 2); purpura (Gr >=2); superior vena cava syndrome (Gr >=1); thromboembolic event (Gr >=2); visceral arterial ischemia (Gr >=2); peripheral arterial ischemia (Gr >=3). TIEs were graded based on Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. For the respective event to count as a treatment-emergent TIE, onset or worsening of the event must have occurred following treatment with PF-05230907 and during the interval between Day 1 dosing through Day 8.
Time Frame: Day 1 through day of discharge (Day 8)
Population: All participants who received the treatment of PF-05230907.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 2

2. Primary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) was any untoward medical occurrence at any dose that: resulted in death; or was life threatening (immediate risk of death); or required inpatient hospitalization or prolongation of existing hospitalization; or resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); or resulted in congenital anomaly/birth defect. Any such events occurring following the start of treatment or increasing in severity were counted as treatment-emergent.
Time Frame: Day 1 through follow-up visit (Day 43)
Population: All participants who received the treatment of PF-05230907.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3
Participants | 0 | 1 | 1 | 0 | 2 | 2

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. For the respective event to count as a treatment-emergent AE, onset or worsening of the event must have occurred following treatment with PF-05230907 and during the interval between Day 1 dosing through Day 8.
Time Frame: Day 1 through day of discharge (Day 8)
Population: All participants who received the treatment of PF-05230907.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3
Participants | 2 | 3 | 3 | 5 | 3 | 3

4. Primary Outcome: Number of Participants With Treatment-Emergent Laboratory Abnormalities
Description: Laboratory safety parameters included hematology, blood chemistry, prothrombin time/international normalized ratio (PT/INR), fibrinogen, antithrombin III (ATIII), Protein S level, Protein C activity, cardiac troponin I, D-dimer, and urinalysis. The number of participants with laboratory test abnormalities meeting specified criteria without regard to baseline abnormality was assessed. Any abnormalities occurring after the administration of treatment and increasing in severity from baseline value were counted as treatment-emergent.
Time Frame: Day 1 through Day 8 (or discharge) for D-dimer laboratory test and urinalysis; Day 1 through Day 4 for all other laboratory tests
Population: All participants who received the treatment of PF-05230907.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3
Participants | 3 | 3 | 3 | 6 | 3 | 3

5. Primary Outcome: Number of Participants With Changes From Baseline in Physical Examination
Description: Comprehensive and targeted physical examinations included general appearance, HEENT (head, eyes, ears, nose and throat), skin, heart (auscultation), lungs (auscultation), abdomen (palpitation and auscultation), and extremities with attention to swelling, general or localized tenderness, entire leg or calf swelling, edema, and collateral superficial veins. The results of the comprehensive and targeted physical examinations were combined to evaluate the changes from baseline through Day 8 (or discharge) for each site parameter according to the categories: positive change (abnormal to normal); no change (normal to normal or abnormal to abnormal); negative change (normal to abnormal). Parameters with at least 1 participant meeting the positive/negative change from baseline criteria are presented here.
Time Frame: Baseline (pre-dose), Day 2, Day 3, Day 4, Day 8/discharge
Population: All participants who received the treatment of PF-05230907.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3
Participants
  Abdomen: Negative change, Day 8/discharge | 0 | 0 | 0 | 1 | 0 | 0
  Extremities: Negative change, Day 2 | 0 | 0 | 0 | 1 | 0 | 0
  Extremities: Negative change, Day 3 | 0 | 0 | 0 | 1 | 0 | 0
  Extremities: Negative change, Day 4 | 0 | 0 | 0 | 1 | 0 | 0
  Extremities: Negative change, Day 8/discharge | 0 | 0 | 0 | 1 | 0 | 0
  Extremities: Positive change, Day 3 | 0 | 0 | 0 | 0 | 0 | 1
  Extremities: Positive change, Day 4 | 0 | 0 | 0 | 0 | 0 | 1
  Extremities: Positive change, Day 8/discharge | 0 | 0 | 0 | 0 | 0 | 1
  Eyes: Negative change, Day 3 | 0 | 0 | 0 | 1 | 0 | 0
  Eyes: Negative change, Day 8/discharge | 0 | 0 | 0 | 1 | 1 | 0
  Eyes: Positive change, Day 2 | 0 | 0 | 0 | 0 | 1 | 0
  Eyes: Positive change, Day 8/discharge | 0 | 0 | 0 | 1 | 1 | 0
  Head: Negative change, Day 2 | 0 | 0 | 0 | 1 | 0 | 0
  Head: Negative change, Day 4 | 0 | 0 | 0 | 1 | 0 | 0
  Head: Positive change, Day 8/discharge | 1 | 0 | 0 | 0 | 0 | 0
  Heart: Negative change, Day 2 | 0 | 0 | 0 | 0 | 1 | 0
  Heart: Negative change, Day 3 | 0 | 0 | 0 | 1 | 0 | 1
  Heart: Negative change, Day 4 | 0 | 0 | 0 | 1 | 0 | 1
  Heart: Negative change, Day 8/discharge | 0 | 0 | 0 | 1 | 0 | 1
  Lungs: Negative change, Day 2 | 0 | 0 | 0 | 0 | 1 | 0
  Lungs: Negative change, Day 4 | 0 | 0 | 0 | 0 | 1 | 0
  Lungs: Negative change, Day 8/discharge | 0 | 0 | 0 | 1 | 1 | 0
  Lungs: Positive change, Day 2 | 0 | 0 | 0 | 0 | 1 | 0
  Lungs: Positive change, Day 8/discharge | 0 | 1 | 0 | 0 | 0 | 1
  Neurological: Negative change, Day 8/discharge | 0 | 0 | 0 | 1 | 0 | 0
  Neurological: Positive change, Day 2 | 0 | 0 | 0 | 0 | 1 | 1
  Neurological: Positive change, Day 3 | 1 | 0 | 0 | 0 | 1 | 0
  Neurological: Positive change, Day 4 | 1 | 0 | 0 | 1 | 2 | 0
  Skin: Positive change, Day 2 | 0 | 0 | 0 | 1 | 0 | 0
  Skin: Positive change, Day 4 | 0 | 0 | 0 | 1 | 0 | 0
  Skin: Positive change, Day 8/discharge | 0 | 0 | 0 | 2 | 0 | 0
  Throat: Negative change, Day 8/discharge | 0 | 0 | 0 | 0 | 1 | 0

6. Primary Outcome: Change From Baseline for Body Temperature
Description: Body temperature was measured by oral, tympanic, axillary or temporal method.
Time Frame: Baseline (pre-dose), Day 1 (5 and 45 minutes [min] post-dose), Day 2, Day 3, Day 4, Day 8/discharge
Population: All participants who received the treatment of PF-05230907. "Number Analyzed" represents the number of participants evaluable for each specified time point.
Measure: Mean (Standard Deviation); unit: Degree Celsius (°C)
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3
Degree Celsius (°C)
  Day 1 (5 min): number analyzed (Participants) | 3 | 3 | 2 | 5 | 3 | 3
  Day 1 (5 min) | 0.1 (0.10) | -0.2 (0.21) | 0.4 (0.57) | -0.1 (0.52) | 0.4 (0.55) | 0.1 (0.10)
  Day 1 (45 min): number analyzed (Participants) | 3 | 3 | 2 | 6 | 3 | 3
  Day 1 (45 min) | 0.1 (0.10) | -0.2 (0.26) | 0.4 (0.57) | -0.1 (0.28) | 0.4 (0.61) | 0.0 (0.30)
  Day 2 | 0.4 (0.76) | 0.5 (0.35) | 0.2 (1.36) | 0.5 (0.98) | 1.0 (1.10) | 0.0 (0.35)
  Day 3 | 0.6 (0.72) | 0.5 (0.20) | 1.1 (0.45) | 1.1 (1.06) | 0.9 (1.63) | 0.1 (0.65)
  Day 4 | 0.1 (0.26) | 0.0 (0.06) | 1.1 (0.99) | 0.4 (0.85) | 0.7 (1.43) | 0.1 (0.25)
  Day 8/discharge: number analyzed (Participants) | 2 | 2 | 3 | 6 | 2 | 3
  Day 8/discharge | -0.2 (0.35) | 0.1 (0.28) | 0.5 (0.70) | 0.4 (0.78) | -0.1 (0.28) | -0.4 (0.68)

7. Primary Outcome: Change From Baseline for Supine Respiratory Rate
Description: Respiratory rate was measured after 5 minutes rest in supine position by observing and counting the respirations of the participant for 30 seconds and multiplied by 2. The use of an automated device for measuring respiratory rate was acceptable.
Time Frame: Baseline (pre-dose), Day 1 (5 and 45 minutes [min] post-dose), Day 2, Day 3, Day 4, Day 8/discharge
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: respiration per minute
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3
respiration per minute
  Day 1 (5 min): number analyzed (Participants) | 3 | 3 | 3 | 4 | 3 | 3
  Day 1 (5 min) | 0.0 (4.00) | 3.7 (3.51) | -1.3 (2.52) | -1.5 (3.00) | -0.3 (0.58) | 0.7 (3.06)
  Day 1 (45 min) | -2.3 (2.08) | 5.7 (1.53) | -0.7 (2.52) | -1.2 (2.93) | 4.0 (6.93) | 0.0 (1.00)
  Day 2 | -1.7 (0.58) | 5.0 (3.61) | -3.0 (1.00) | -0.8 (2.86) | 0.0 (2.00) | -0.7 (0.58)
  Day 3 | -1.0 (3.00) | 5.3 (2.89) | -1.0 (2.65) | 0.0 (4.15) | 1.7 (2.89) | 0.3 (2.52)
  Day 4 | 0.3 (2.52) | 4.0 (3.46) | -0.7 (3.79) | -1.0 (2.19) | 1.3 (4.16) | -0.7 (1.15)
  Day 8/discharge: number analyzed (Participants) | 2 | 2 | 3 | 6 | 2 | 3
  Day 8/discharge | -2.5 (0.71) | 2.5 (0.71) | -2.0 (2.65) | 1.2 (2.71) | -1.0 (1.41) | -2.7 (2.89)

8. Primary Outcome: Change From Baseline for Supine Systolic and Diastolic Blood Pressure
Description: Supine blood pressure (BP, systolic and diastolic) was measured with the participant's arm supported at the level of the heart and recorded to the nearest milliliters of mercury (mmHg) after 5 minutes of rest whenever possible and as permitted by the participant's medical condition.
Time Frame: Baseline (pre-dose), Day 1 (5 and 45 minutes [min] post-dose), Day 2, Day 3, Day 4, Day 8/discharge
Population: All participants who received the treatment of PF-05230907. "Number Analyzed" represents the number of participants evaluable for each specified category.
Measure: Mean (Standard Deviation); unit: milliliters of mercury (mmHg)
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3
milliliters of mercury (mmHg)
  Supine Systolic BP, Day 1 (5 min): number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 3
  Supine Systolic BP, Day 1 (5 min) | -6.3 (13.28) | 27.7 (27.65) | -4.3 (8.14) | -10.2 (12.56) | 11.0 (12.12) | 9.7 (7.23)
  Supine Systolic BP, Day 1 (45 min) | -13.3 (12.01) | 15.0 (36.76) | -5.3 (38.28) | -26.7 (27.53) | 12.0 (20.95) | -6.7 (29.54)
  Supine Systolic BP, Day 2 | -3.3 (8.14) | -7.3 (17.01) | -11.0 (11.53) | -29.8 (25.63) | -14.0 (8.54) | 0.7 (18.58)
  Supine Systolic BP, Day 3 | -14.3 (19.09) | 5.3 (17.93) | 12.0 (7.21) | -36.2 (26.16) | 5.3 (34.56) | -15.7 (3.79)
  Supine Systolic BP, Day 4 | -12.0 (17.09) | 6.3 (30.37) | -6.0 (12.49) | -32.5 (25.84) | 7.3 (11.93) | -27.7 (17.21)
  Supine Systolic BP, Day 8/discharge: number analyzed (Participants) | 2 | 2 | 3 | 6 | 2 | 3
  Supine Systolic BP, Day 8/discharge | -18.0 (5.66) | -1.0 (26.87) | -5.0 (18.03) | -22.8 (50.01) | 18.5 (3.54) | -14.3 (6.35)
  Supine Diastolic BP, Day 1 (5 min): number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 3
  Supine Diastolic BP, Day 1 (5 min) | -9.0 (15.59) | 10.7 (11.02) | -7.3 (15.53) | -21.6 (20.94) | 5.3 (9.24) | 6.3 (2.08)
  Supine Diastolic BP, Day 1 (45 min) | -11.3 (17.62) | 7.3 (21.83) | 9.3 (1.15) | -27.0 (25.11) | 1.7 (7.64) | 2.0 (2.65)
  Supine Diastolic BP, Day 2 | -0.7 (12.06) | -8.0 (4.00) | -4.7 (21.73) | -26.2 (32.39) | -7.3 (1.53) | -5.7 (8.74)
  Supine Diastolic BP, Day 3 | -7.0 (6.24) | -4.3 (11.93) | 5.0 (8.66) | -28.2 (24.81) | 4.0 (12.17) | -6.7 (4.16)
  Supine Diastolic BP, Day 4 | -14.0 (10.58) | -8.3 (16.17) | 8.7 (17.67) | -26.5 (21.77) | -5.7 (12.06) | -11.0 (19.97)
  Supine Diastolic BP, Day 8/discharge: number analyzed (Participants) | 2 | 2 | 3 | 6 | 2 | 3
  Supine Diastolic BP, Day 8/discharge | -12.0 (2.83) | -4.0 (11.31) | 12.0 (19.67) | -24.2 (36.31) | 2.5 (7.78) | -6.0 (6.24)

9. Primary Outcome: Change From Baseline for Supine Pulse Rate
Description: The use of an automated device for measuring pulse rate was acceptable, although, when done manually, pulse rate was measured in the brachial/radial artery for at least 30 seconds.
Time Frame: Baseline (pre-dose), Day 1 (5 and 45 minutes [min] post-dose), Day 2, Day 3, Day 4, Day 8/discharge
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3
beats per minute (bpm)
  Day 1 (5 min): number analyzed (Participants) | 3 | 3 | 3 | 4 | 3 | 3
  Day 1 (5 min) | -0.7 (5.69) | 1.3 (4.16) | 1.7 (1.53) | 0.0 (2.45) | -17.3 (17.01) | 2.7 (4.62)
  Day 1 (45 min) | 8.0 (20.07) | -1.3 (23.18) | -2.7 (7.51) | -0.2 (5.98) | -13.3 (10.07) | 2.7 (14.19)
  Day 2 | -13.0 (19.97) | -21.0 (18.73) | 5.7 (1.15) | -2.7 (5.89) | -11.0 (16.37) | -3.3 (21.50)
  Day 3 | -12.3 (22.28) | -13.0 (7.94) | 1.0 (12.00) | 9.2 (13.53) | -14.3 (17.21) | 3.0 (25.94)
  Day 4 | -13.7 (31.53) | -21.0 (12.12) | -11.0 (9.85) | -3.7 (10.84) | -12.7 (30.17) | 7.3 (18.77)
  Day 8/discharge: number analyzed (Participants) | 2 | 2 | 3 | 6 | 2 | 3
  Day 8/discharge | -16.5 (36.06) | -18.0 (7.07) | -1.7 (4.16) | 6.2 (8.04) | -34.0 (0.00) | 2.0 (5.57)

10. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Qualitative Results
Description: The electrocardiogram (ECG) results over time were compared to baseline and assessed by the investigator as "less abnormal", "no significant change", or "more abnormal".
Time Frame: Baseline (pre-dose), Day 2, Day 4, Day 8/discharge
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3
Participants
  Day 2: Less abnormal | 0 | 0 | 0 | 0 | 0 | 0
  Day 2: No significant change | 3 | 3 | 3 | 6 | 3 | 3
  Day 2: More abnormal | 0 | 0 | 0 | 0 | 0 | 0
  Day 4: number analyzed (Participants) | 3 | 3 | 3 | 6 | 2 | 3
  Day 4: Less abnormal | 0 | 0 | 0 | 0 | 0 | 0
  Day 4: No significant change | 3 | 3 | 3 | 6 | 2 | 2
  Day 4: More abnormal | 0 | 0 | 0 | 0 | 0 | 1
  Day 8/discharge: number analyzed (Participants) | 2 | 2 | 3 | 6 | 2 | 3
  Day 8/discharge: Less abnormal | 0 | 0 | 0 | 2 | 0 | 0
  Day 8/discharge: No significant change | 2 | 2 | 3 | 4 | 2 | 2
  Day 8/discharge: More abnormal | 0 | 0 | 0 | 0 | 0 | 1

11. Secondary Outcome: Maximum Changes From Baseline for Activated Partial Thromboplastin Time (aPTT)
Description: Maximum changes from baseline were calculated for activated partial thromboplastin time (aPTT) after dosing with PF-05230907 through Day 2.
Time Frame: Baseline (pre-dose), Day 2
Population: All treated participants who had at least 1 measurement of pharmacodynamic parameters of interest.
Measure: Mean (Standard Deviation); unit: seconds (sec)
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3
seconds (sec) | -8.53 (3.250) | -12.17 (1.060) | -8.47 (1.790) | -8.76 (4.859) | -5.00 (5.522) | -12.03 (4.574)

12. Secondary Outcome: Maximum Changes From Baseline for Prothrombin Fragment 1+2 (PF1+2)
Description: Maximum changes from baseline were calculated for prothrombin fragment 1+2 (PF1+2) after dosing with PF-05230907 through Day 2.
Time Frame: Baseline (pre-dose), Day 2
Population: All treated participants who had at least 1 measurement of pharmacodynamic parameters of interest.
Measure: Mean (Standard Deviation); unit: picomoles per liter (pmol/L)
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3
picomoles per liter (pmol/L) | -163.7 (390.08) | 2823.7 (137.25) | 1286.0 (1331.09) | 492.6 (1445.60) | 1773.7 (1472.95) | 354.3 (501.75)

13. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) Production
Description: Participants with anti-drug antibody (ADA) production were those with at least 1 positive result from Day 1 through follow-up visit (Day 43 and/or Day 91). ADA positive: titer value >=1.88.
Time Frame: Day 1 up to follow-up visit (Day 43 and/or Day 91)
Population: All treated participants who had at least 1 measurement of post-treatment immunogenicity parameters of interest.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Neutralizing Antibody (NAb) Production
Description: ADA positive samples were planned to be further characterized for neutralizing antibody (NAb). Participants with NAb production were those with at least 1 positive result from Day 1 through follow-up visit (Day 43 and/or Day 91). As all ADA samples were negative (titer value <1.88), NAb analysis was not conducted.
Time Frame: Day 1 up to follow-up visit (Day 43 and/or Day 91)
Population: All treated participants who had at least 1 measurement of post-treatment immunogenicity parameters of interest.
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Depletion of Coagulation Factor X
Description: Depletion of coagulation factor X was defined as >50% reduction relative to baseline (pre-dose).
Time Frame: Baseline (pre-dose), Day 43, Day 91
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3
Participants
  Day 43: number analyzed (Participants) | 3 | 3 | 2 | 4 | 2 | 2
  Day 43 | 0 | 0 | 0 | 0 | 0 | 0
  Day 91: number analyzed (Participants) | 2 | 1 | 2 | 4 | 1 | 1
  Day 91 | 0 | 0 | 0 | 0 | 0 | 0

16. Other Pre Specified Outcome: Change From Baseline in Intracerebral Hemorrhage (ICH) Volume at 24 Hours
Description: Change from baseline in intracerebral hemorrhage (ICH) volume was calculated at 24 hours.
Time Frame: Baseline (pre-dose), 24 hours
Population: All participants who received the treatment of PF-05230907.
Measure: Mean (Standard Deviation); unit: centimeter (cm)^3
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3
centimeter (cm)^3 | -0.297 (0.3761) | 0.410 (2.1554) | 12.137 (10.9207) | 1.190 (2.1099) | 1.130 (1.7385) | 0.097 (1.8781)

17. Other Pre Specified Outcome: PF-05230907 Concentration in Plasma
Time Frame: Day 1 pre-dose, 5 and 45 minutes post-dose
Population: All treated participants who had at least 1 measurement of PF-05230907 concentration. "Number Analyzed" represents the number of participants evaluable for each specified category.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3
nanogram per milliliter (ng/mL)
  Pre-dose: number analyzed (Participants) | 3 | 2 | 3 | 5 | 3 | 3
  Pre-dose | NA (NA) — Mean and standard deviation (SD) were not available as none of the analyzed participants had plasma PF-05230907 concentration above the lower limit of quantification (LLOQ). The LLOQ was 1.95 ng/mL. | NA (NA) — Mean and SD were not available as none of the analyzed participants had plasma PF-05230907 concentration above the LLOQ. The LLOQ was 1.95 ng/mL. | 17.46 (28.121) | 2.382 (3.4180) | NA (NA) — Mean and SD were not available as none of the analyzed participants had plasma PF-05230907 concentration above the LLOQ. The LLOQ was 1.95 ng/mL. | NA (NA) — Mean and SD were not available as none of the analyzed participants had plasma PF-05230907 concentration above the LLOQ. The LLOQ was 1.95 ng/mL.
  5 minutes post-dose: number analyzed (Participants) | 3 | 0 | 3 | 5 | 2 | 3
  5 minutes post-dose | 11.90 (13.359) |  | 34.63 (30.731) | 39.82 (28.393) | 35.60 (21.072) | 41.17 (23.756)
  45 minutes post-dose: number analyzed (Participants) | 3 | 2 | 3 | 4 | 1 | 3
  45 minutes post-dose | 1.377 (1.1935) | 2.460 (0.32527) | 17.21 (23.815) | 6.938 (1.6070) | 2.490 (NA) — SD was not available as only 1 participant was analyzed. | 4.657 (1.6342)

18. Other Pre Specified Outcome: Number of Participants With Anti-Chinese Hamster Ovary (CHO) Protein Antibody Production
Description: Participants with anti-Chinese hamster ovary (CHO) antibody production were those with positive results. Positive: titer value >=2.00.
Time Frame: Day 1, Day 43
Population: All treated participants who had at least 1 measurement of post-treatment immunogenicity parameters of interest. "Number Analyzed" represents the number of participants evaluable for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3
Participants
  Day 1: number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 2
  Day 1 | 0 | 1 | 2 | 2 | 2 | 1
  Day 43: number analyzed (Participants) | 3 | 3 | 2 | 4 | 2 | 2
  Day 43 | 0 | 1 | 2 | 3 | 2 | 2

19. Other Pre Specified Outcome: Number of Participants With Anti-Paired Basic Amino Acid Cleaving Enzyme (PACE) Furin Antibody Production
Description: Participants with anti-paired basic amino acid cleaving enzyme (PACE) antibody production were those with positive results. Positive: titer value >=2.00.
Time Frame: Day 1, Day 43
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3
Participants
  Day 1 | 0 | 0 | 0 | 0 | 0 | 0
  Day 43: number analyzed (Participants) | 3 | 3 | 2 | 4 | 2 | 2
  Day 43 | 0 | 0 | 0 | 0 | 0 | 0

20. Other Pre Specified Outcome: Neurological Function as Assessed by the National Institute of Health Stroke Scale (NIHSS)
Description: The National Institute of Health Stroke Scale (NIHSS) is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. The total NIHSS score range is from 0 (normal) to 42 (severe impairment), with higher values indicating greater level of neurological impairment.
Time Frame: Screening, Day 1, Day 2, Day 4, Day 43, and Day 91
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3
units on a scale
  Screening | 11.7 (7.37) | 10.7 (8.62) | 15.3 (10.60) | 15.7 (4.68) | 17.0 (2.65) | 13.7 (7.51)
  Day 1: number analyzed (Participants) | 3 | 3 | 3 | 6 | 2 | 3
  Day 1 | 11.3 (6.81) | 14.0 (6.24) | 15.3 (10.60) | 15.2 (6.37) | 16.0 (2.83) | 13.7 (7.51)
  Day 2: number analyzed (Participants) | 2 | 3 | 3 | 6 | 2 | 3
  Day 2 | 10.0 (12.73) | 16.3 (6.51) | 16.0 (10.82) | 12.3 (5.43) | 16.0 (4.24) | 14.3 (5.86)
  Day 4: number analyzed (Participants) | 3 | 3 | 3 | 6 | 2 | 3
  Day 4 | 5.7 (8.08) | 12.7 (8.14) | 16.0 (10.82) | 9.8 (5.98) | 13.5 (2.12) | 14.7 (6.03)
  Day 43: number analyzed (Participants) | 3 | 3 | 2 | 5 | 2 | 2
  Day 43 | 1.0 (1.00) | 8.3 (8.39) | 4.5 (6.36) | 4.4 (5.59) | 15.5 (4.95) | 5.0 (1.41)
  Day 91: number analyzed (Participants) | 3 | 2 | 2 | 5 | 2 | 2
  Day 91 | 0.7 (0.58) | 1.5 (0.71) | 3.5 (3.54) | 5.2 (5.07) | 13.5 (7.78) | 2.0 (2.83)

21. Other Pre Specified Outcome: Health Resource Utilization Surrogate Measures - Maximum Duration
Description: Maximum duration for 4 types of hospital or health care unit: Intensive Care Unit (ICU), general ward, rehabilitation center, and other hospital units. This was an exploratory endpoint to evaluate information for designing future studies, which were no longer planned.
Time Frame: Day 1 up to Day 91
Population: as for outcome 8
Measure: Median (Full Range); unit: days
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3
days
  ICU: number analyzed (Participants) | 1 | 1 | 1 | 2 | 2 | 1
  ICU | 2 [NA to NA] — NA as only 1 participant had data. | 2 [NA to NA] — NA as only 1 participant had data. | 1 [NA to NA] — NA as only 1 participant had data. | 30 [1 to 59] | 17.5 [4 to 31] | 1 [NA to NA] — NA as only 1 participant had data.
  General ward: number analyzed (Participants) | 1 | 3 | 2 | 3 | 2 | 3
  General ward | 1 [NA to NA] — NA as only 1 participant had data. | 5 [1 to 7] | 16.5 [16 to 17] | 7 [6 to 7] | 31.5 [0 to 63] | 26 [5 to 42]
  Rehabilitation center: number analyzed (Participants) | 1 | 3 | 2 | 4 | 1 | 2
  Rehabilitation center | 75 [NA to NA] — NA as only 1 participant had data. | 75 [61 to 79] | 40.5 [22 to 59] | 30.5 [26 to 43] | 79 [NA to NA] — NA as only 1 participant had data. | 20 [14 to 26]
  Other hospital unit: number analyzed (Participants) | 2 | 2 | 1 | 2 | 2 | 0
  Other hospital unit | 4 [4 to 4] | 3 [2 to 4] | 7 [NA to NA] — NA as only 1 participant had data. | 24 [17 to 31] | 3.5 [1 to 6] |

ADVERSE EVENTS:
Time Frame: For each participant, Adverse Events (AEs) were collected up to Day 43/follow-up visit. All-Cause Mortality table presents all deaths up to 3.4 months.
Description: An AE may be categorized as serious in 1 participant and as non-serious in another participant; 1 participant may have experienced both a serious and non-serious AE.
Arm/Group | PF-05230907 5 Microgram Per Kilogram (mcg/kg) | PF-05230907 8 mcg/kg | PF-05230907 12 mcg/kg | PF-05230907 19 mcg/kg | PF-05230907 24 mcg/kg | PF-05230907 30 mcg/kg
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 1/3 | 0/6 | 2/3 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 1/3 | 0/6 | 2/3 | 2/3
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 3/3 | 5/6 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-05230907 5 Microgram Per Kilogram (mcg/kg) (N=3) | PF-05230907 8 mcg/kg (N=3) | PF-05230907 12 mcg/kg (N=3) | PF-05230907 19 mcg/kg (N=6) | PF-05230907 24 mcg/kg (N=3) | PF-05230907 30 mcg/kg (N=3)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Stroke in evolution (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-05230907 5 Microgram Per Kilogram (mcg/kg) (N=3) | PF-05230907 8 mcg/kg (N=3) | PF-05230907 12 mcg/kg (N=3) | PF-05230907 19 mcg/kg (N=6) | PF-05230907 24 mcg/kg (N=3) | PF-05230907 30 mcg/kg (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site phlebitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain management (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated after 21 participants were enrolled for a strategic reason, not for safety nor efficacy reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-01-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT02687191/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT02687191/SAP_001.pdf